CLINICAL TRIAL: NCT03913676
Title: Disseminating a Waitlist Treatment for Anxiety With Velibra
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not feasible.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jasper A. Smits, Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-11-0128
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Velibra (Experimental): All treatment will be provided via the Velibra website: https://velibra.broca.io/en/registration/voucher. While the Velibra treatment is only six weeks long, participants will have free access to the program for 24 weeks. They can access this website as often as they would like. The Velibra program is self-guided, so participants determine how often they access the material (the program encourages participants to complete one of six sessions per week for six weeks).
  Interventions: Behavioral: Velibra

INTERVENTIONS:
Behavioral: Velibra — Velibra is grounded in a cognitive-behavioral theoretical orientation and consists of six treatment modules representing different skills and therapeutic techniques. Each of the first five modules is followed by a "training session", and contains activities related to training attention biases (CBM-I). All sessions plus trainings are designed to be completed in 1 - 2 hours, depending on the user's reading speed, interest, motivation, and individual path through the program. The modules cover a variety of therapeutic content that is broadly consistent with a cognitive-behavioral perspective. The modules' content draws from therapeutic strategies: (1) Cognitive Modification, (2) Mindfulness, Acceptance, and Relaxation techniques (4) Exposure, (5) Interpersonal Skills, (6) Psychoeducation and Relapse Prevention.

SUMMARY:
Cognitive Behavioral Therapy (CBT) is a gold standard treatment for a wide spectrum of anxiety-related concerns. However, long waitlist times can serve as a substantial barrier to those seeking treatment. Internet delivered psychotherapy, such as internet-based CBT (I-CBT) may present an affordable option for disseminating empirically supported treatments. Velibra, an web-based I-CBT intervention, has shown initial promise in treating anxiety disorders.

Velibra has been used to treat anxiety-related disorders in European samples with participants recruited from general practitioner's offices and diagnosed with a specific subset of anxiety disorders. While these effects are encouraging, additional research is needed toevaluate whether Velibra could be implemented in a community mental health clinic in the U.S. Specifically, if Velibra could be successfully implemented within the context of mental health clinic waitlists, it may be capable of providing evidence-based treatment to larger groups of people at a faster rate than mental health clinics can structurally support.

The purpose of this study is to assess the feasibility of implementing Velibra into an American community clinic waitlist. We plan to offer free access to the Velibra program to members of the Anxiety and Stress Clinic (ASC) waitlist at the University of Texas at Austin experiencing anxiety. We will evaluate interest in the program, user data from the program, and opinions of the program post-completion. We hypothesize ASC patients will find utility in Velibra's ability to offer them mental health resources faster than the traditional waitlist can provide.

DETAILED DESCRIPTION:
Waitlist Recruitment. Participants will be recruited directly from the Anxiety and Stress Clinic's waitlist. Consistent with our existing clinic screening procedures, individuals added to our waitlist meeting the following criteria will be invited to participate in this study:

1. They have not experienced significant suicidal ideation in the past week.
2. They do not meet for a bipolar I diagnosis without current utilization of stabilizing medications.
3. They are not experiencing psychotic symptoms.

Upon meeting these criteria and being added to the clinic waitlist, patients will be asked if they would like to participate in our feasibility trial. Patients already on the waitlist at the time of study approval will also be contacted and offered participation. If interested in participating, patients will be asked to complete a digital informed consent via UT Qualtrics or Research Electronic Data Capture (REDCap), secure, online assessment tools designed to collect self-report questionnaire data for research studies.

Baseline Survey. Following informed consent, participants will complete a baseline survey via UT Qualtrics or REDCap. This survey will include measures of anxiety and other internalizing symptoms (Patient Health Questionnaire, PHQ-9; Generalized Anxiety Disorder 7-item Scale, GAD-7; Overall Anxiety Severity and Impairment Scale, OASIS). Other questions will evaluate participants' current medication/treatment status (Treatment/Medication Status questions). More details about these questionnaires included below. Following completion of the baseline survey, participants will receive a voucher for free access to Velibra.

Velibra Program. All treatment will be provided via the Velibra website: https://velibra.broca.io/en/registration/voucher. While the Velibra treatment is only six weeks long, participants will have free access to the program for 24 weeks. They can access this website as often as they would like. The Velibra program is self-guided, so participants determine how often they access the material (the program encourages participants to complete one of six sessions per week for six weeks).

Velibra Treatment. Velibra is grounded in a cognitive-behavioral theoretical orientation and consists of six treatment modules representing different skills and therapeutic techniques. Each of the first five modules is followed by a "training session", and contains activities related to training attention biases (CBM-I). All sessions plus trainings are designed to be completed in 1 - 2 hours, depending on the user's reading speed, interest, motivation, and individual path through the program. Modules are organized as simulated dialogues in which the program explains and illustrates concepts and techniques, engages the user in exercises, and continuously asks users to respond by selecting from response options. Subsequent content is then tailored to the users' responses, resulting in a simulated conversational flow. All modules are accompanied by illustrations (e.g., drawings, photographs, flash animations). The modules cover a variety of therapeutic content that is broadly consistent with a cognitive-behavioral perspective, although the program is not restricted to one CBT manual. Instead, the program provides a variety of relevant therapeutic approaches and fits within the broad array of contemporary CBT. The modules' theoretical rationale and content draws from therapeutic strategies: (1) Cognitive Modification, (2) Mindfulness, Acceptance, and Relaxation techniques (4) Exposure, (5) Interpersonal Skills, (6) Psychoeducation and Relapse Prevention.

Throughout participants' use of the program, we will collect user data on Velibra's secure, online server (amount of time spent in the program, number of completed modules, number of training sessions completed between modules).

Post-Treatment Survey. Six weeks after the original voucher send date, participants will be asked to complete a second survey via UT Qualtrics or REDCap. This survey will include identical symptom measures (PHQ-9; GAD-7; OASIS) and will contain a series of questions about Anxiety and Stress Clinic treatment interest and Velibra dropout (Participation Questions). Lastly, the survey will include questions about current medication/treatment status (Treatment/Medication Status Questions) as well as questions concerning user satisfaction (SUS), credibility of treatment (CSQ-8), and other questions for suggestions (Suggestions).

ELIGIBILITY:
Inclusion Criteria:

* Currently on the Anxiety and Stress Clinic waitlist
* At least 18 years old
* Fluent in English
* Have access to a computer or web device

Exclusion Criteria:

* Active suicidal ideation with intent to harm oneself in the past week (e.g., endorses "Yes" toC-SSRS item 4 or higher).
* A formal diagnosis of Bipolar I disorder without current utilization of stabilizing medications.
* Present or past psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Feasibility (Percentage of participants who complete at least one module) | [assessed at 6-week follow-up]
  Percentage of participants who complete at least one module of Velibra (out of the total number of participants offered access to the program).

SECONDARY OUTCOMES:
System Usability Scale (Brooke, 1996) | [assessed at 6-week follow-up]
  Measures quality of a program's interface; final scores determined by summing all 10-items of self-report scale, with higher totals reflecting higher interface quality; minimum score = 10; maximum score = 50
Client Satisfaction Questionnaire (Larsen, Attkisson, Hargreaves, & Nguyen, 1979) | [assessed at 6-week follow-up]
  Measures participant satisfaction with the program; final scores determined by summing all 8-items of self-report scale, with higher totals reflecting higher satisfaction with the program; minimum score = 8; maximum score = 32
Treatment-Seeking Behavior | [assessed at 6-week follow-up]
  Percentage of participants who would like to enroll in traditional CBT treatment at 6 week follow-up (out of the total number of participants who completed at least one module of Velibra).
Overall Anxiety Severity and Impairment Scale (Norman, Hammi Cissell, Means-Christensen, & Stein, 2006) | [assessed at baseline and 6-week follow-up]
  Measures anxiety symptoms and impact on functioning; final scores determined by summing all 5-items of self-report scale, with higher totals reflecting larger levels of anxiety symptoms; minimum score = 0; maximum score = 20
Generalized Anxiety Disorder Scale-7 (Spitzer, Kroenke, Williams, & Lowe, 2006) | [assessed at baseline and 6-week follow-up]
  Measures anxiety symptoms; final scores determined by summing all 7-items of self-report scale, with higher totals reflecting larger levels of anxiety symptoms; minimum score = 0; maximum score = 21
Patient Health Questionnaire (Kroenke, Spitzer, & Williams, 2001) | [assessed at baseline and 6-week follow-up]
  Measures depressive symptoms; final scores determined by summing all 9-items of self-report scale, with higher totals reflecting larger levels of depressive symptoms; minimum score = 0; maximum score = 27

CONTACTS AND LOCATIONS:
Overall Officials: Jasper A.J. Smits, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berger T, Urech A, Krieger T, Stolz T, Schulz A, Vincent A, Moser CT, Moritz S, Meyer B. Effects of a transdiagnostic unguided Internet intervention ('velibra') for anxiety disorders in primary care: results of a randomized controlled trial. Psychol Med. 2017 Jan;47(1):67-80. doi: 10.1017/S0033291716002270. Epub 2016 Sep 22. PMID 27655039
- [Background] Brooke, J. (1996). SUS-A quick and dirty usability scale. Usability Evaluation in Industry, 189(194), 4-7.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Norman SB, Cissell SH, Means-Christensen AJ, Stein MB. Development and validation of an Overall Anxiety Severity And Impairment Scale (OASIS). Depress Anxiety. 2006;23(4):245-9. doi: 10.1002/da.20182. PMID 16688739
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Priester MA, Browne T, Iachini A, Clone S, DeHart D, Seay KD. Treatment Access Barriers and Disparities Among Individuals with Co-Occurring Mental Health and Substance Use Disorders: An Integrative Literature Review. J Subst Abuse Treat. 2016 Feb;61:47-59. doi: 10.1016/j.jsat.2015.09.006. Epub 2015 Oct 31. PMID 26531892
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Hofmann SG, Smits JA. Cognitive-behavioral therapy for adult anxiety disorders: a meta-analysis of randomized placebo-controlled trials. J Clin Psychiatry. 2008 Apr;69(4):621-32. doi: 10.4088/jcp.v69n0415. PMID 18363421